CLINICAL TRIAL: NCT02918656
Title: Presenting Summary Information From Cochrane Systematic Reviews: Randomized Controlled Trial of Infographics Presentation vs. Standard Word Summaries
Brief Title: Presenting Summary Information From Cochrane Systematic Reviews
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Split (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Ivan Buljan, PhD student, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IP-2014-09-7672
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Understanding Cochrane Systematic Reviews
Keywords: Cochrane; Abstract; Infographics; Understanding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Infographics (Experimental): Infographic presentation of health information
  Interventions: Other: Infographic presentation of health information
- Plain Language Summary (Active Comparator): PLS presentation of health information
  Interventions: Other: PLS presentation of health information
- Scientific abstract (Active Comparator): Scientific abstract presentation of health information
  Interventions: Other: Scientific abstract presentation of health information

INTERVENTIONS:
Other: Infographic presentation of health information — The students in this group will read Cochrane systematic review summary in infographics format.
  Infographics format is a form of visual presentation of results of systematic review, supported by pictures and graphs.
  Arms: Infographics
Other: PLS presentation of health information — The students randomized in PLS group will read text format with simple explanation of the survey topic main findings which is intended for lay audience.
  Arms: Plain Language Summary
Other: Scientific abstract presentation of health information — The students in scientific abstract group will read the the text written for the academic population and practitioners.
  Arms: Scientific abstract

SUMMARY:
The objective of the investigators study is to evaluate the efficacy of infographics in presenting information, in terms of understanding and remembering research results, compared to standard PLS formats and scientific summary formats (SciSum).

DETAILED DESCRIPTION:
The investigators will conduct a randomized control trial (RCT) with three different formats of the same systematic review summary (infographics, PLS and scientific summary). The content of these three formats is based on the same systematic review, but the ways of data presentation will differ: visual presentation, plain language, and scientific language. The trial will be performed at the beginning of the 2016/2017 academic year, with first year university students as participants. The trial will be voluntary and anonymous. The survey will consist of 4 parts: 1) demographic data, 2) one format of the summary (randomly assigned), 3) comprehension test of the information given in the summary, 4) accessibility of information and overall satisfaction with the given summary assessed by survey and 5) health numeracy test. All materials will be in Croatian. The materials used in this research will be assessed by experts in order to confirm face validity of developed questions.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be first-year university students without experience with Cochrane review summaries, because prior familiarization with Cochrane summaries could make information uptake easier by those participants.

Exclusion criteria:

* Participants who give the positive answer to the survey question about familiarity with the Cochrane will be excluded from the study analysis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2016-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Marušić, MD, PhD, Principal Investigator — Professor at Medical School of Split
Locations (1):
- School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: No
Data will be collected electronically, using the SurveyMonkey platform. The data will be fully anonymous and will be kept on a secure server of the School of Medicine.

RESULTS

PARTICIPANT FLOW:
Groups:
- Infographics: Infographic presentation of health information
  Infographic presentation of health information: The students in this group will read Cochrane systematic review summary in infographics format.
  Infographics format is a form of visual presentation of results of systematic review, supported by pictures and graphs.
Period: Overall Study
Arm/Group | Infographics | Plain Language Summary | Scientific Abstract
Started | 54 | 60 | 57
Completed | 54 | 60 | 57
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infographics | Plain Language Summary | Scientific Abstract | Total
Number analyzed (Participants) | 54 | 60 | 57 | 171
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 19 [19 to 21] | 19 [19 to 20] | 19 [19 to 21] | 19 [19 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 50 | 142
  Male | 10 | 12 | 7 | 29
Heard of Cochrane systematic reviews [Count of Participants; unit: Participants] | 5 | 2 | 2 | 9
Used Cochrane library [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Primary source of health information [Count of Participants; unit: Participants]
  Internet | 25 | 31 | 29 | 85
  Family Members | 15 | 11 | 15 | 41
  Family physician | 11 | 16 | 11 | 38
  Library | 2 | 2 | 2 | 6
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Understanding
Description: The primary outcome of the study is the score on a understanding test with ten questions about information contained in all three forms of presentation, titled as "Understanding information about external cephalic version for breech presentation before term" (Hutton et al, 2015). The questions will focus on understanding the benefits and risks of the intervention and the quality of evidence described in the systematic review. Each correctly answered question will be awarded one point, with a maximum of 10 points. The scale was specifically designed for this research, they ask about the information contained in all three abstract format and all questions are open-ended.
Time Frame: One-hour after the intervention
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Infographics | Plain Language Summary | Scientific Abstract
Number analyzed (Participants) | 54 | 60 | 57
units on a scale | 6.0 [5.0 to 7.0] | 6.0 [5.1 to 6.0] | 5.0 [4.0 to 5.0]

2. Secondary Outcome: Reading Experience
Description: This section of the survey will include 5 questions about the experience of participants about the text they read, measured on a 10-point Likert type scale, where 1 means do not agree at all and 10 means fully agree. The total score is the sum of scores on all five answers (minimum score was 10 and maximum 50). Higher scores indicate greater reading experience, which means that a person was assessed that type of reading material as more enjoyable. So, higher scores are associated with more positive reading experience.
Time Frame: One hour after the intervention
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Infographics | Plain Language Summary | Scientific Abstract
Number analyzed (Participants) | 54 | 60 | 57
units on a scale | 31.0 [27.8 to 33.0] | 30 [26.1 to 32.0] | 16.0 [14.3 to 18.0]

3. Secondary Outcome: Accessibility of Relevant Information
Description: This section of the survey will have 5 questions concerning how easy it was for the participant to find relevant information, measured by a 10-point Likert type scale where the answer 1 means I do not agree at all and 10 means I fully agree. The total score is the sum of scores on all the answers (minimum score was 5, maximum 50). The higher score indicated that the reading material was perceived as more user friendly and that it was easier to find the desired information.
Time Frame: One hour after the intervention
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Infographics | Plain Language Summary | Scientific Abstract
Number analyzed (Participants) | 54 | 60 | 57
units on a scale | 32.5 [30.0 to 34.5] | 32.5 [31.0 to 35.0] | 19.5 [17.0 to 21.0]

4. Secondary Outcome: Health Numeracy Score
Description: This section will use 6-item General health numeracy test (Osborne et al., 2013) in order to determine how much our participants understand the basic health instructions regarding numeracy dimension. For each correct answer, the participants receive one point and the total score is the sum of all correct answers.
Time Frame: One hour after the intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Infographics | Plain Language Summary | Scientific Abstract
Number analyzed (Participants) | 54 | 60 | 57
units on a scale | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.8] | 3.0 [2.0 to 4.0]

ADVERSE EVENTS:
Time Frame: Adverse events data was not collected.
Description: 0
Arm/Group | Infographics | Plain Language Summary | Scientific Abstract
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor had no role in planning of research, its execution nor publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT02918656/Prot_SAP_000.pdf